CLINICAL TRIAL: NCT02213250
Title: An Open-label, Single Dose Pharmacokinetic Study Of Benefix (Nonacog Alfa, Recombinant Factor Ix) In Male Chinese Subjects With Hemophilia B
Brief Title: An Open-Label, Single Dose Pharmacokinetic Study of Benefix (Recombinant Factor IX) in Male Chinese Subjects With Hemophilia B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1821048; 2015-003027-61 (EudraCT Number)
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Results first posted 2016-07-25 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-06

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B | interventions — Factor IX

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BeneFIX (Experimental)
  Interventions: Drug: BENEFIX

INTERVENTIONS:
Drug: BENEFIX — Single dose of 50 IU/kg of BeneFIX by intravenous infusion within 10 minutes.

SUMMARY:
The sample size of 12 male Chinese subjects are based on the CFDA requirement for a China PK study and to support the registration in China.

ELIGIBILITY:
Inclusion Criteria:

* Male Chinese subjects 6 years or older (weight ≥20kg) with moderate to severe hemophilia B (Factor IX activity ≤2%).
* Subjects should not have received an infusion of any Factor IX products for at least 4 days before the administration of BeneFIX on Day 1.
* Subjects must be in a non-bleeding state before the administration of BeneFIX on Day 1.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) disease or clinical findings at Screening.
* Diagnosed with any other bleeding disorder in addition to hemophilia B.
* Current FIX inhibitor or history of FIX inhibitor (defined as > Upper Limit of Normal (ULN) of the reporting lab).

Min Age: 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- China (2):
  - Peking Union Medical College Hospital, Beijing
  - Hematology Department,Beijing Children's Hospital, Capital Medical University, Beijing

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1821048&StudyName=An%20Open-Label%2C%20Single%20Dose%20Pharmacokinetic%20Study%20of%20Benefix%20%28Recombinant%20Factor%20IX%29%20in%20Male%20Chinese%20Subjects%20with%20Hemophilia%20B%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twelve (12) participants that were age 6 years or older (weight ≥20 kg) with moderate severe to severe hemophilia B (FIX activity ≤2%) were enrolled. Four (4) participants were at the younger age range of ≥6 and <12 years; remaining participants were 12 years or older.
Pre-assignment Details: Participants did not receive an infusion of any FIX products for at least 4 days and were required to be in a non-bleeding state before the administration of BeneFIX on Day 1.
Groups:
- BeneFIX 50 IU/kg; Age Group: >=6 and <12 Years: Participants received a single dose of 50 IU/kg BeneFIX administered by intravenous (IV) infusion within 10 minutes at approximately 0800 hours (±2 hours) on Day 1.
- BeneFIX 50 IU/kg; Age Group: >=12 Years: Participants received a single dose of 50 IU/kg BeneFIX administered by IV infusion within 10 minutes at approximately 0800 hours (±2 hours) on Day 1.
Period: Overall Study
Arm/Group | BeneFIX 50 IU/kg; Age Group: >=6 and <12 Years | BeneFIX 50 IU/kg; Age Group: >=12 Years
Started | 4 | 8
Completed | 4 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants were included in the baseline population.
Groups:
- All Participants: Participants received a single dose of 50 IU/kg BeneFIX administered by IV infusion within 10 minutes at approximately 0800 hours (±2 hours) on Day 1.
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 24.8 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Pre-dose, 0.25, 0.5, 1, 3, 6, 9, 24, 50, 72 and 96 hours post-dose
Population: The pharmacokinetics (PK) parameter analysis population was defined as all participants enrolled and treated who had at least 1 of the PK parameters of primary interest. All participants were included in the PK analysis population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/milliliter (IU/mL)
Groups:
- BeneFIX 50 IU/kg; >=6 and <12 Years; BeneFIX 50 IU/kg; Age Group:>=12 Years: Participants received a single dose of 50 IU/kg BeneFIX administered by IV infusion within 10 minutes at approximately 0800 hours (±2 hours) on Day 1.
Arm/Group | BeneFIX 50 IU/kg; >=6 and <12 Years | BeneFIX 50 IU/kg; Age Group:>=12 Years
Number analyzed (Participants) | 4 | 8
IU/milliliter (IU/mL) | 0.3880 (26) | 0.4226 (16)

2. Primary Outcome: Area Under the Concentration Time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUClast)
Time Frame: Pre-dose, 0.25, 0.5, 1, 3, 6, 9, 24, 50, 72 and 96 hours post-dose
Population: The PK parameter analysis population was defined as all participants enrolled and treated who had at least 1 of the PK parameters of primary interest. All participants were included in the PK analysis population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU*hour/milliliter (IU*hr/mL)
Arm/Group | BeneFIX 50 IU/kg; >=6 and <12 Years | BeneFIX 50 IU/kg; Age Group:>=12 Years
Number analyzed (Participants) | 4 | 8
IU*hour/milliliter (IU*hr/mL) | 6.930 (18) | 9.707 (15)

3. Primary Outcome: Area Under the Concentration Time Curve From Time 0 to Infinity (AUCinf)
Time Frame: Pre-dose, 0.25, 0.5, 1, 3, 6, 9, 24, 50, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU*hr/ml
Groups:
- BeneFIX 50 IU/kg; Age Group>=6 and <12 Years; BeneFIX 50 IU/kg; Age Group:>=12 Years: Participants received a single dose of 50 IU/kg BeneFIX administered by IV infusion within 10 minutes at approximately 0800 hours (±2 hours) on Day 1.
Arm/Group | BeneFIX 50 IU/kg; Age Group>=6 and <12 Years | BeneFIX 50 IU/kg; Age Group:>=12 Years
Number analyzed (Participants) | 4 | 8
IU*hr/ml | 7.841 (16) | 11.66 (15)

4. Primary Outcome: Time to Reach Cmax (Tmax)
Time Frame: Pre-dose, 0.25, 0.5, 1, 3, 6, 9, 24, 50, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | BeneFIX 50 IU/kg; >=6 and <12 Years | BeneFIX 50 IU/kg; Age Group:>=12 Years
Number analyzed (Participants) | 4 | 8
hours | 0.500 [0.250 to 3.00] | 0.375 [0.250 to 3.00]

5. Primary Outcome: Volume of Distribution at Steady State (Vss)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Vss is the apparent volume of distribution at steady-state.
Time Frame: Pre-dose, 0.25, 0.5, 1, 3, 6, 9, 24, 50, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter/kilogram (mL/kg)
Arm/Group | BeneFIX 50 IU/kg; >=6 and <12 Years | BeneFIX 50 IU/kg; Age Group:>=12 Years
Number analyzed (Participants) | 4 | 8
milliliter/kilogram (mL/kg) | 227.9 (20) | 218.8 (19)

6. Primary Outcome: Terminal Phase Rate Constant (Kel)
Description: Linear regression of the log linear concentration time curve. Only those data points judged to describe the terminal log linear decline were used in the regression.
Time Frame: Pre-dose, 0.25, 0.5, 1, 3, 6, 9, 24, 50, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hr
Arm/Group | BeneFIX 50 IU/kg; >=6 and <12 Years | BeneFIX 50 IU/kg; Age Group:>=12 Years
Number analyzed (Participants) | 4 | 8
1/hr | 0.02509 (16) | 0.01781 (20)

7. Primary Outcome: Mean Residence Time (MRT)
Description: AUMCinf/AUCinf, where AUMCinf is the area under the first moment curve from time 0 extrapolated to infinite time, calculated using the linear/log trapezoidal method.
Time Frame: Pre-dose, 0.25, 0.5, 1, 3, 6, 9, 24, 50, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | BeneFIX 50 IU/kg; >=6 and <12 Years | BeneFIX 50 IU/kg; Age Group:>=12 Years
Number analyzed (Participants) | 4 | 8
hours | 35.78 (14) | 51.01 (16)

8. Primary Outcome: Plasma Decay Half-Life (t½)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Pre-dose, 0.25, 0.5, 1, 3, 6, 9, 24, 50, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BeneFIX 50 IU/kg; >=6 and <12 Years | BeneFIX 50 IU/kg; Age Group:>=12 Years
Number analyzed (Participants) | 4 | 8
hours | 27.88 (4.4903) | 39.56 (7.3832)

9. Primary Outcome: Systemic Clearance (CL)
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: Pre-dose, 0.25, 0.5, 1, 3, 6, 9, 24, 50, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hr/kg
Arm/Group | BeneFIX 50 IU/kg; >=6 and <12 Years | BeneFIX 50 IU/kg; Age Group:>=12 Years
Number analyzed (Participants) | 4 | 8
mL/hr/kg | 6.378 (16) | 4.291 (15)

10. Primary Outcome: Incremental Recovery
Description: Incremental recovery: Increase in circulating increase in FIX activity for every IU of BeneFIX administered per kg of body weight.
Time Frame: Pre-dose, 0.25, 0.5 and 1 hour post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (IU/dL)/(IU/Kg)
Arm/Group | BeneFIX 50 IU/kg; >=6 and <12 Years | BeneFIX 50 IU/kg; Age Group:>=12 Years
Number analyzed (Participants) | 4 | 8
(IU/dL)/(IU/Kg) | 0.7759 (26) | 0.8199 (17)

11. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAE), Serious Adverse Events (SAE), and Withdrawals Due to Adverse Events (AE)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; lifethreatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. TEAE is defined as newly occurring or worsening after first dose.
Time Frame: From the subject provided informed consent through and including 28 calendar days after the last administration of the study drug.
Population: The safety analysis set was defined as all participants who received at least 1 dose of BeneFIX.
Measure: Number; unit: Particpants
Groups:
- BeneFIX 50 IU/kg: Participants received a single dose of 50 IU/kg BeneFIX administered by IV infusion within 10 minutes at approximately 0800 hours (±2 hours) on Day 1.
Arm/Group | BeneFIX 50 IU/kg
Number analyzed (Participants) | 12
Particpants | 0

12. Secondary Outcome: Number of Participants With Abnormal Clinical Laboratory Measurements (Without Regard to Baseline Abnormality)
Description: Clinical laboratory analysis tests included hematology, serium chemistry, prothrombin time and urianalysis. Numbers of subjects with laboratory test abnormalities without regard to baseline abnormality were reported.
Time Frame: Baseline up to 96 hours post-dose (Day 5 or early termination)
Population: The safety analysis population included All participants who received at least 1 dose of BeneFIX.
Measure: Number; unit: Participants
Arm/Group | BeneFIX 50 IU/kg
Number analyzed (Participants) | 12
Participants | 12

13. Secondary Outcome: Number of Participants With Vital Signs Post-Dose Data Met Criteria of Potential Clinical Concern (Without Regard to Baseline Abnormality)
Time Frame: Baseline up to 96 hours post-dose (Day 5 or early termination)
Population: The safety analysis population included All participants who received at least 1 dose of BeneFIX.
Measure: Number; unit: Participants
Arm/Group | BeneFIX 50 IU/kg
Number analyzed (Participants) | 12
Participants | 1

14. Secondary Outcome: Number of Participants With Inhibitor Development
Time Frame: as for outcome 11
Population: The safety analysis population included All participants who received at least 1 dose of BeneFIX.
Measure: Number; unit: Participants
Arm/Group | BeneFIX 50 IU/kg
Number analyzed (Participants) | 12
Participants | 0

15. Secondary Outcome: Number of Participants With Allergic Reactions
Time Frame: as for outcome 11
Population: The safety analysis population included All participants who received at least 1 dose of BeneFIX.
Measure: Number; unit: Participants
Arm/Group | BeneFIX 50 IU/kg
Number analyzed (Participants) | 12
Participants | 0

16. Secondary Outcome: Number of Subjects With Thrombogenicity
Time Frame: as for outcome 11
Population: The safety analysis population included All participants who received at least 1 dose of BeneFIX.
Measure: Number; unit: Participants
Arm/Group | BeneFIX 50 IU/kg
Number analyzed (Participants) | 12
Participants | 0

ADVERSE EVENTS:
Time Frame: From the subject provided informed consent through and including 28 calendar days after the last administration of the study drug.
Arm/Group | BeneFIX 50 IU/kg
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restriction Description: Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.